CLINICAL TRIAL: NCT05804799
Title: Comparison of Image Quality and Diagnostic Pefromance of Low Dose Liver CT With Deep Learning Reconstuction to Standard Dose CT: A Prospective Multicenter Non-inferiority Trial
Brief Title: Liver CT Dose Reduction With Deep Learning Based Reconstruction
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: SNUH-2007-040-1139
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Radiation Exposure; Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Liver CT study group: Patients with a suspicion of focal liver lesions had the plan to perform a contrast-enhanced liver CT scan.
  The liver CT images were reconstructed by both low-dose scans with a deep-learning-based denoising program (ClariCT.AI) and standard-dose scans with model-based iterative reconstruction.
  Interventions: Diagnostic Test: Contrast-enhanced liver CT scan

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced liver CT scan — The contrast-enhanced liver CT scans were obtained from all of the participants.
  The liver CT images were reconstructed by both low-dose scans with a deep-learning-based denoising program (ClariCT.AI) and standard-dose scans with model-based iterative reconstruction.

SUMMARY:
A deep learning-based de-noising (DLD) reconstruction algorithm (ClariCT.AI) has the potential to reduce image noise and improve image quality. This capability of the CliriCT.AI program might enable dose reduction for contrast-enhanced liver CT examination. In this prospective multicenter study, whether the ClariCT.AI program can reduce the noise level of low-dose contrast-enhanced liver CT (LDCT) data and therefore, can provide comparable image quality to the standard dose of contrast-enhanced liver CT (SDCT) images will be evaluated.

The aim of this study is to compare image quality and diagnostic capability in detecting malignant tumors of LDCT with DLD to those of SDCT with MBIR using the predefined non-inferiority margin.

DETAILED DESCRIPTION:
A deep learning-based de-noising (DLD) reconstruction algorithm (ClariCT.AI) has the potential to reduce image noise and improve image quality. This capability of the CliriCT.AI program might enable dose reduction for contrast-enhanced liver CT examination. In this prospective multicenter study, whether the ClariCT.AI program can reduce the noise level of low-dose contrast-enhanced liver CT (LDCT) data and therefore, can provide comparable image quality to the standard dose of contrast-enhanced liver CT (SDCT) images will be evaluated.

The aim of this study is to compare image quality and diagnostic capability in detecting malignant tumors of LDCT with DLD to those of SDCT with MBIR using the predefined non-inferiority margin.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-year-old and 85 years old
* patients referred to the Radiology department to perform contrast-enhanced liver CT under the suspicion of focal liver lesions

Exclusion Criteria:

* patients with estimated glomerular filtration rate < 60 mL/min/1.73m2
* previous history of severe adverse reaction to iodinated contrast media.

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a suspicion of focal liver lesions had the plan to do a contrast-enhanced liver CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of standard deviation of CT attenuation values at the liver | within 6 months from acquisition of liver CT scans
  Standard deviation of CT attenuation values at the liver parenchyma

SECONDARY OUTCOMES:
Sensitivity to detect malignant liver tumor | within 6 months from acquisition of liver CT scans
  Sensitivity of liver CT scans to detect malignant liver tumor

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (3):
- Tubingen University Hospital, Tübingen, Germany
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee DH, Lee JM, Lee CH, Afat S, Othman A. Image Quality and Diagnostic Performance of Low-Dose Liver CT with Deep Learning Reconstruction versus Standard-Dose CT. Radiol Artif Intell. 2024 Mar;6(2):e230192. doi: 10.1148/ryai.230192. PMID 38231025